CLINICAL TRIAL: NCT02153463
Title: Enhancing Physical Activity in Children With Tics and Tourette Syndrome: Impact on Tic Severity and Quality of Life
Brief Title: Activity in Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Asif Doja, Assistant Professor, Associate Investigator, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14/72X
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Tourette Syndrome; Persistent Tic Disorder
Keywords: Tourette Syndrome; Persistent Tic Disorder; Physical Activity; Quality of Life
MeSH Terms: conditions — Tourette Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activity Counselling (Experimental): Physical Activity Counselling weekly for 8 weeks
  Interventions: Behavioral: Physical Activity Counselling
- Standard Care (No Intervention): Standard care with no change in medications for 8 weeks

INTERVENTIONS:
Behavioral: Physical Activity Counselling — Physical Activity Counselling weekly for 8 weeks
  Arms: Activity Counselling

SUMMARY:
Tics are brief repetitive movements or vocalizations. Gilles de la Tourette's syndrome (TS) is a disorder characterized by recurrent motor and vocal tics. Tourette syndrome and tic disorders affect up to 8% of children. Peak severity of tic disorders occurs between the ages of 8 to 12 years, therefore during childhood and adolescence the most significant impacts are felt. The quality of life of young people with tics is lower than their peers' and tic severity predicts lower quality of life. Studies have also shown negative social perception toward children with tics.

Approximately 50% of patients with Tourette syndrome will have other diagnoses including attention deficit hyperactivity disorder (ADHD), obsessive compulsive disorder, anxiety and depression. Studies have shown improvements in ADHD with physical activity. ADHD and tic disorders are thought to involve the same areas of the brain; thus it is possible that tics might also improve with physical activity. However, no studies to date have examined this. The investigators predict that by implementing a motivational physical activity program, in conjunction with physical activity counseling, the investigators will be able to increase levels of physical activity in children with tics and Tourette syndrome, with a positive impact on tic severity.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between 8-16 years of age.
* Participants are required to have a diagnosis of either Tourette Syndrome or Persistent (Chronic) Motor of Vocal Tic Disorder as per the DSM V.
* Participants must be ambulatory.
* Participants and parents must understand English or French.
* Participants must be able and willing to complete the questionnaires.
* Participants cannot have any changes to their medication for tics, or any other psychotropic medications for 4 weeks prior to and for the entire duration of the study

Exclusion Criteria:

* Participants who cannot ambulate independently.
* Participants who are not permitted to participate in physical education class at school.
* Participants or families who are not willing to be randomly assigned to a study group.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Decrease in Yale Global Tic Severity Scale. | 8 weeks

SECONDARY OUTCOMES:
Change in The Gilles de la Tourette Syndrome Quality of Life Scale for children and adolescents | 8 weeks

OTHER OUTCOMES:
Change in PedsQL 4.0 measure | 8 weeks
Change in KidScreen-27 | 8 weeks
Chang in The Children's Self-perceived Adequacy and Predilection for Physical Activity Questionnaire | 8 Weeks
Change in step count via pedometer | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Doja A, Bookwala A, Pohl D, Rossi-Ricci A, Barrowman N, Chan J, Longmuir PE. Relationship Between Physical Activity, Tic Severity and Quality of Life in Children with Tourette Syndrome. J Can Acad Child Adolesc Psychiatry. 2018 Nov;27(4):222-227. Epub 2018 Nov 1. PMID 30487937